CLINICAL TRIAL: NCT03120663
Title: Target Attainment and Pharmacokinetics of Antimicrobials in Non-critically Ill Surgery Patients
Brief Title: Target Attainment and Pharmacokinetics of Antimicrobials in Non-critically Ill Surgery Patients (TAPAS)
Acronym: TAPAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, peter declercq, Principal investigator, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S59726
Record Dates: First submitted 2017-04-04; First posted 2017-04-19 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Surgery
Keywords: antimicrobials; pharmacokinetics; augmented renal clearance; non critically ill
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination; Meropenem; Floxacillin; Piperacillin, Tazobactam Drug Combination; Clindamycin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Per patient, blood samples during 1 antimicrobial dosing interval and the measured creatinine clearance based on an 8-hour urinary collection (CrCl8h) will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: amoxicillin-clavulanic acid — During one dosing interval at steady state of the involved antimicrobials (ABs), AB plasma concentrations will be determined.
  Besides, the measured creatinine clearance based on an 8-hour urinary collection (CrCl8h) will be used as the primary method for determining kidney function. Based on these values, CrCl8h will be calculated according to the standard formula and normalized to a body surface area (BSA) of 1.73m² .
  Other Names: meropenem; flucloxacillin; piperacillin-tazobactam; clindamycin

SUMMARY:
In this prospective observational study, the investigators want to document pharmacokinetic/pharmacodynamic (PK/PD) target attainment of frequently used antimicrobials in an adult non critically ill surgery population (abdominal surgery, traumatology and septic orthopedic surgery). Furthermore, the investigators want to identify risk factors for not attaining predefined PK/PD targets.

The antibiotics of interest are amoxicillin(-clavulanic acid), flucloxacillin, piperacillin-tazobactam, meropenem and clindamycin.

DETAILED DESCRIPTION:
In this research proposal, the primary objective is to describe PK parameters (area under the curve (AUC), clearance (Cl), distribution volume (Vd) and half life (T1/2)) for the antibiotics of interest (amoxicillin(-(clavulanic acid), flucloxacillin, piperacillin-tazobactam, meropenem and clindamycin) for this adult non critically ill surgery population.

Besides, the investigators want to document pharmacokinetic/pharmacodynamic (PK/PD) target attainment of frequently used ABs in this population and to identify risk factors, for example augmented renal clearance (ARC), for not attaining predefined PK/PD targets.

ELIGIBILITY:
Inclusion Criteria:

Every adult non-critically ill surgery patient admitted at the abdominal, trauma or septic orthopaedic surgery wards from the University Hospitals Leuven treated with multiple doses of one of the antimicrobials of interest (i.e. intravenous (IV) amoxicillin(-clavulanic acid), flucloxacillin, piperacillin-tazobactam, meropenem, oral or IV clindamycin) is eligible for inclusion.

Exclusion Criteria:

* age ≤ 18 years
* treatment restrictions corresponding to a Do Not Reanimate code
* pregnancy
* lactation
* renal replacement therapy
* planned discharge or surgery in the coming antimicrobial dosing interval making sampling impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult non-critically ill surgery patient admitted at the abdominal, trauma or septic orthopaedic surgery wards from the University Hospitals Leuven
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-11-30 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
The % of time that free concentrations of antimicrobials are above minimal inhibitory concentrations (MIC) or antimicrobial European Committee on Antimicrobial Susceptibility Testing (EUCAST) breakpoints | During 1 dosing interval at steady state. This is at earliest 72h after initialization of the antimicrobial.
  Per antimicrobial of interest, we will determine the % of time that free concentrations are above minimal inhibitory concentrations (MIC) or antimicrobial EUCAST breakpoints

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | During 1 dosing interval at steady state. This is at earliest 72h after initialization of the antimicrobial.
  Per antimicrobial of interest, we will determine the pharmacokinetic parameter the area under the plasma concentration versus time curve (AUC).
Clearance (Cl) | During 1 dosing interval at steady state. This is at earliest 72h after initialization of the antimicrobial.
  Per antimicrobial of interest, we will determine the pharmacokinetic parameter clearance (Cl).
Volume of distribution (Vd) | During 1 dosing interval at steady state. This is at earliest 72h after initialization of the antimicrobial.
  Per antimicrobial of interest, we will determine the pharmacokinetic parameter the volume of distribution (Vd).
Half life (T1/2) | During 1 dosing interval at steady state. This is at earliest 72h after initialization of the antimicrobial.
  Per antimicrobial of interest, we will determine the pharmacokinetic parameter the half life (T1/2).
Risk factors for target non attainment | During 1 dosing interval at steady state. This is at earliest 72h after initialization of the antimicrobial.
  Multivariate analysis will be performed with target attainment as outcome. This will allow to identify risk factors for target non attainment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Declercq, PharmD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No